CLINICAL TRIAL: NCT00430703
Title: Effect of Massive Proprioceptive Stimulation With Passive Gait Training on the Cortical Activity in Patients With Impaired States of Consciousness After Severe Traumatic Brain Injury.
Brief Title: Effect of Passive Gait Training on the Cortical Activity in Patients With Severe Traumatic Brain Injury.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus County, Denmark (Other)
Responsible Party: Natallia Lapitskaya, MD, Hammel Neurorehabilitation and Research Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNRC-AAU-06-1
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Craniocerebral Trauma; Traumatic Brain Injury; "Rehabilitation"
Keywords: severe traumatic brain injury; body weight support treadmill training; Electroencephalogram; Event Related Potentials
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients with severe traumatic brain injury
  Interventions: Behavioral: body weight support treadmill training
- 2 (Experimental): Healthy volunteers
  Interventions: Behavioral: body weight support treadmill training

INTERVENTIONS:
Behavioral: body weight support treadmill training — Gait training: Gait robot (Lokomat®, Hocoma, Switzerland) is adjusted to the patient/healthy volunteer individually with chest strap, pelvic straps, harness, leg cuffs and foot lifters. Weight is adjusted individually, so there is a minimum weight support (i.e. when one foot is standing on the treadmill the other foot lifts free from the treadmill thereby simulating normal gait). Gait speed is 1,7-2,3 km/hour (speed can be changed and adjusted that the normal step length is achieved).The duration of the training session is 20 minutes.Blood pressure and pulse are monitored.

SUMMARY:
The aim of this study is to determine whether passive gait training increases arousal, demonstrated as changes in EEG (electroencephalogram) activity.

Hypotheses: 1) Passive gait training increases EEG-frequency in patients with impaired consciousness due to severe traumatic brain injury.

2) Passive gait training increases conductivity speed of the cognitive P300-component of ERP in patients with impaired consciousness due to severe traumatic brain injury.

DETAILED DESCRIPTION:
Severe traumatic brain injury, especially after a high energy trauma, is characterised with focal lesions and diffuse axonal injury, which leads to the dysfunction in the cortico-spinal, cortico- cortical connections and reticular activation system. Formatio reticularis plays an important role in arousal. Tactile and proprioceptive stimulation with a view to improving level of consciousness in coma patients is popular in the western world despite insufficient evidence of its effectiveness. Affolter-Bobath-Coombes-concept is the most commonly used tool in the rehabilitation of brain damaged patients. This concept is based on the theory that tactile, proprioceptive and oral stimulation develops new connections in the brain and thereby stimulates consciousness and behaviour. Elliot et al shows improvement in level of consciousness due to postural changes from a lying position to a standing posture in 8 of 12 patients using Wessex Head Injury Matrix.

Passive movements result in proprioceptive stimulation; the effect of which is close to that achieved by physiological voluntary activity. PET and fMRI studies show that passive movements activate several areas in the motor cortex.

In order to increase afferent cortical input, passive gait training in the body weight support robotic gait orthosis could be used in patients with impaired consciousness, inability to cooperate and poor balance. This device gives the possibility to establish therapeutically correct upright body position and passive legs movement simultaneously.

To our knowledge there are no studies, which illustrate the effects of passive gait training on cortical activity in patients with impaired consciousness due to severe traumatic brain injury.

Our hypothesis is that passive gait training of this group of patients increases arousal, which can be shown in an increased EEG (electroencephalogram)-frequency and increased conductivity speed of the cognitive P300-component of ERP (Event Related Potentials).

Comparison(s): EEG- and ERP-activity after a single training session in robotic gait orthosis in patients with severe traumatic brain injury, compared to EEG- and ERP-activity after a single training session in robotic gait orthosis in healthy persons.

ELIGIBILITY:
Inclusion Criteria:

Patient group :

1. severe brain injury (GCS-scale< 8 on admission to the hospital);
2. Ongoing impaired state of consciousness (RLAS-scale≤4);
3. stable vital functions;
4. written consent from relatives/ legal guardian.

Control group:

1. no history of neurological diseases in the past;
2. age over 18 years;
3. written agreement.

Exclusion Criteria:

Patient and control group:

1. age older than 80 years;
2. other neurological disease;
3. lack of BAEP and SEP;
4. severe co-morbidity;
5. pregnancy;
6. robotic orthosis contraindications (orthostatic circulatory problems, unstable fractures, severe osteoporosis, skin problems, joint problems, severe asymmetry (major difference in leg length over 2 cm), co-operation problems (reduced cooperation, psychotic illnesses or neurotic disturbances), body weight over 100 kg, adjustment problems (i.e. robot cannot be safely adjusted to the patient).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
EEG: difference in the frequency spectrum after training. | 0-30 minutes after training end

SECONDARY OUTCOMES:
EEG: absolute power i every frequency band; median frequency; | 0-30 minutes after training end
frequency ratios: Alpha versus delta;delta and theta versus alpha and beta; | 0-30 minutes after training end
ERP: amplitude of P300-component. | 30-60 minutes after training end
ERP: latency of P300-component. | 30-60 minutes after training
clinical measure: RLAS (Rancho Los Amigos Scale) | discharge from the rehabilitation unit

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Koch-Jensen, MD, Study Director — Hammel Neurorehabilitation and Research Centre; Johannes Jakobsen, MD, DMSc, Study Chair — Department of Neurology, Aarhus University; Natallia Lapitskaya, MD, PhD-stud, Principal Investigator — Hammel Neurorehabilitation and Research Centre
Locations (1):
- Hammel Neurorehabilitation and Research Centre, Hammel, Denmark